CLINICAL TRIAL: NCT03356522
Title: TRIFIR : Study of Trabecular Bone Score (TBS) as a Fracture Risk Factor in Chronic Renal Failure
Brief Title: Study of Trabecular Bone Score (TBS) as a Fracture Risk Factor in Chronic Renal Failure
Acronym: TRIFIR
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3029_TRIFIR
Record Dates: First submitted 2017-11-16; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Chronic Renal Failure; Kidney Transplant Patients
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study

DETAILED DESCRIPTION:
The Trabecular Bone Score (TBS) is a recent imaging tool that indirectly studies bone microarchitecture from 2-dimensional images of lumbar biphotonic absorptiometry (DXA). His interest is demonstrated in the evaluation of the fracture risk of the general population. The study of its interest in chronic renal failure is ongoing, only 3 studies have been published to our knowledge.

Osteopathy of chronic renal failure is a complex phenomenon involving bone remodeling disorders, mineralization, mass and bone microarchitecture. In the renal transplant population, certain factors, such as anti-rejection therapy, are also involved.

The impact of fragility fractures induced by these disorders of bone metabolism is a major public health issue due to the resulting morbidity and mortality, with mortality doubling in comparison to the general population after a hip fracture.

The bone osteopathy assessment of chronic renal failure is the bone biopsy, however its realization is very limited because of its invasiveness.

Although initially Bone Densitometry was not recommended in the evaluation of the fracture risk of chronic renal failure by KDIGO (Kidney Disease Improvement Global Outcomes) of 2009, many works published since plead in favor of its realization for the fracture risk assessment, in combination with the clinical data of the Fracture Risk Assessment Tool (FRAX), as should be recommended in the next KDIGO. Indeed, the decrease in bone density in chronic renal failure is associated with an increased risk of fracture.

Clinical parameters, of course, also play an important role in the evaluation of the fracture risk of chronic renal insufficiency, be it the items taken into account in FRAX, certain factors related to chronic kidney disease, or even transplantation. kidney transplant.

To our knowledge, only three studies on the association of TBS with fracture risk of chronic renal failure have been published. In particular, they show a significant association between the decrease in TBS and the incident fracture risk, independently of bone density and FRAX, in a population of kidney transplant recipients, and chronic renal insufficiency in stage 3 or 4.

According to KDIGO 2009, the only biomarkers recommended in the evaluation of osteopathy chronic renal failure are parathyroid hormone (PTH) and bone-specific alkaline phosphatase (BAP), although there is no established threshold for significant increase in fracture risk . However, there is little data on other bone remodeling markers such as the Procollagen type 1 N-terminal propeptide (P1NP) and the C-terminal telopeptide of type 1 collagen (CTX). Some studies indicate, however, that they may be of interest in evaluation of osteopathy of chronic renal failure .

ELIGIBILITY:
Inclusion Criteria:

* 1st population: kidney failure patients at stage 4-5, age> 40 years, non-dialyzed, ungrafted.
* 2nd population: kidney transplant patients, age> 40, first kidney transplant.

Exclusion Criteria:

* Pregnant women.
* Incapable adults (tutelage, guardianship, safeguard of justice).
* Persons deprived of liberty.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney failure patients and kidney transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Value of Trabecular Bone Score (TBS) | Baseline

SECONDARY OUTCOMES:
Evaluation of bone remodeling markers | Baseline
  Biological markers: parathyroid hormone (PTH)
Evaluation of bone remodeling markers | Baseline
  Biological markers: Bone-specific Alkaline Phosphatase (BAP)
Evaluation of bone remodeling markers | Baseline
  Biological markers: Procollagen type 1 N-terminal propeptide (P1NP)
Evaluation of bone remodeling markers | Baseline
  Biological markers: C-terminal telopeptide of type I collagen (CTX)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Guggenbuhl, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Britain, France